CLINICAL TRIAL: NCT04460118
Title: Clinical and Radiographic Outcomes in Arthroscopic "Inlay"Bristow Surgery With Screw Fixation vs Suture-button Fixation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: cui1
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Shoulder; Dislocation, Chronic
MeSH Terms: conditions — Joint Dislocations; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- screw group: coracoid bone block fixed by the screw
  Interventions: Procedure: Bristow surgery fixed by the screw
- button group: coracoid bone block fixed by the suture-button
  Interventions: Procedure: Bristow surgery fixed by the suture button

INTERVENTIONS:
Procedure: Bristow surgery fixed by the screw — Bristow surgery fixed by the screw
  Groups: screw group
Procedure: Bristow surgery fixed by the suture button — Bristow surgery fixed by the suture button
  Groups: button group

SUMMARY:
Retrospective comparative case-cohort study to investigate the efficacy of the modified arthroscopic Bristow-Latarjet surgery and to compare the clinical and radiographic outcomes using screw fixation vs suture-button fixation.

DETAILED DESCRIPTION:
Background：Some studies have advocated the use of suture-button fixation during Bristow-latarjet surgery to reduce complications associated with screw fixation. However, these studies are not comparative studies, and their data are relatively incomplete.

Purpose: To compare the clinical and radiographic outcomes using screw fixation vs suture-button fixation.

Study Design: Retrospective comparative case-cohort study Methods: Patients who underwent the modified arthroscopic Bristow-Latarjet surgery between June 2015 and February 2018 were selected. Shoulders were separated into two groups based on surgical fixation method. Radiological results on 3D CT scan and clinical results were assessed preoperatively, immediately after operation, and postoperatively at 3 months, 6 months, 1 year and during the final follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. a glenoid defect ≥10%
2. contact sport athletes with a glenoid defect < 10%
3. failure after Bankart repair.

Exclusion Criteria:

1. epilepsy
2. multidirectional shoulder instability
3. concomitant other lesions including rotator cuff tear, symptomatic acromioclavicular joint pathology or pathological involvement of the long head of the biceps
4. Follow-up was less than 2 years or incomplete follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients undergoing the "Inlay" Bristow surgery in our hospital between June 2015 and February 2018.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
VAS for pain score | 2 years after surgery
  The visual analog scale (VAS) for pain score is the most commonly used to describe pain levels in patients, ranging from 0 to 10, with a higher score indicating more intense pain.
ASES score | 2 years after surgery
  The American Shoulder and Elbow Surgeons (ASES) score is the most commonly used score to describe the function of patients' shoulder joints, ranging from 0 to 100. The higher the score, the better the function of patients' shoulder joints.

SECONDARY OUTCOMES:
Active shoulder ranges of motion | 2 years after surgery
  internal rotation at the side, and external and internal rotation at 90° of abduction,
Bone block position | immediately after surgery.
  Bone block position was evaluated using postoperative CT scans.The ideal position of the bone block was defined as flush to the anterior glenoid rim in the axial view and 4 o'clock in the En face view. The bone block was considered too lateral if it went beyond the glenoid rim by more than 5 mm and it was judged to be too medial if it was medial to the rim by more than 5 mm.
Bone union | 3 months after surgery, 6 months after surgery, 1 year after surgery and 2 years after surgery
  Graft union with the glenoid was assessed using postoperative CT scans. ''Bony union'' of the transplant was defined as no radiolucent zone; ''fibrous union,'' when the transplant had a radiolucent zone of less than 5 mm; and ''migration,'' when the zone was 5 mm or more.

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, professor, Principal Investigator — Peking University Third Hospital
Locations (1):
- PekingUTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No